CLINICAL TRIAL: NCT00735358
Title: Comparison of Endoscopic Injection of Conventional and Double Doses Cyanoacrylate for Gastric Variceal Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Chan Cho-Yu, M.D, / excutive officer of IRB of Taipei VGH, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95DHA0100359
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2008-08

CONDITIONS: Gastric Variceal Bleeding
Keywords: gastric variceal bleeding; cyanoacrylate; rebleeding; complication; survival; acute gastric variceal bleeding
MeSH Terms: interventions — Cyanoacrylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Single dose cyanoacrylate in one shot
  Interventions: Procedure: Cyanoacrylate
- B (Experimental): Double doses cyanoacrylate in one shot
  Interventions: Procedure: Cyanoacrylate

INTERVENTIONS:
Procedure: Cyanoacrylate — Cyanoacrylate 0.5 ml, endoscopic injection of gastric varix at each shot
  Arms: A
Procedure: Cyanoacrylate — Cyanoacrylate 1 ml, endoscopic injection for gastric varices at each shot
  Arms: B

SUMMARY:
The recent practice guideline recommends endoscopic injection of cyanoacrylate (GVO) is the preferred method to treat acute gastric variceal bleeding. The rebleeding rate remains high following GVO.We hypothesized that a double-dose of cyanoacrylate may obliterate the varices more effectively and achieve better hemostasis.

DETAILED DESCRIPTION:
Although outcome of variceal hemorrhage has been improved in the last two decades, variceal hemorrhage is still the most serious complication of portal hypertension and chronic liver disease. Occurrence of gastric varices (GV) rupture is less often than esophageal varices (EV) but it is characteristic of higher rebleeding rate and mortality and represents an even tougher problem than EV hemorrhage. Facing these challenges, there is no consensus on the best treatment of GV hemorrhage and therefore it is mainly empirical. Endoscopic treatment is an alternative in the management of GVH. Injection sclerotherapy has been applied to arrest GV hemorrhage but it is associated with a high rebleeding rate (50~90%) and thus is regarded as only a temporary hemostatic measure. The advantage of endoscopic variceal ligation for EV hemorrhage has been documented, however, endoscopic variceal ligation for GVH is not as promising because of its high rebleeding rate around 50%. Endoscopic injection of N-butyl-2-cyanoacrylate, a so-called "tissue glue", was more effective for GV hemorrhage than other sclerosants and endoscopic ligation, however, its rebleeding rate is still high around 30~50%. The theoretical advantages of tissue glue derives from its unique ability to plug the varix lumen immediately. Each injection of tissue glue in conventional use was usually prepared by a mixture of 0.5 ml cyanoacrylate and 0.5 ml Lipiodol. Therefore, we hypothesized that double dose cyanoacrylate (1 ml cyanoacrylate mixed with 1 ml Lipiodal) may obliterate the varices in further distance and broader area and that may achieve more effective hemostatic results than conventional dose. Therefore we designed a randomized trial to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis and/or hepatoma
* Aged 18 to 80, who had endoscopy-proven acute GVB
* Clinical signs of hematemesis, coffee ground vomitus, hematochezia, or melena
* Endoscopic signs of active bleeding from the GV
* Adherent blood clots, white nipple signs, or erosions on the GV
* The presence of distinct large GV with red-color signs and absence of EV and other bleeding sources
* Who or their legally authorized representatives gave informed consent

Exclusion Criteria:

* Patients had previous endoscopic, surgical treatment or transjugular intrahepatic portosystemic shunt (TIPS) for GVB
* Had a terminal illness of any major organ system, such as heart failure, uremia, chronic pulmonary disease, or non-hepatic malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Rebleeding | 2 year

SECONDARY OUTCOMES:
Survival | 2 year

REFERENCES:
- [Derived] Hou MC, Lin HC, Lee HS, Liao WC, Lee FY, Lee SD. A randomized trial of endoscopic cyanoacrylate injection for acute gastric variceal bleeding: 0.5 mL versus 1.0 mL. Gastrointest Endosc. 2009 Oct;70(4):668-75. doi: 10.1016/j.gie.2009.02.005. Epub 2009 Jun 25. PMID 19559427